CLINICAL TRIAL: NCT06736106
Title: ORTHOSPINE FITNESS: Which Markers of Musculoskeletal Health Can Explain Complications in Spinal Surgery?
Brief Title: Which Markers of Musculoskeletal Health Can Explain Complications in Spinal Surgery?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: Azienda Ospedaliera Universitaria Luigi Vanvitelli (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OrthoSpine Fitness; PNRR-MCNT2-2023-12378098 (Other Grant/Funding Number: Ministero della Salute.)
Record Dates: First submitted 2024-12-06; First posted 2024-12-16 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Spine Injuries and Disorders
Keywords: spine surgery; muscle strength; physical fragility; musculoskeletal system; degenerative pathologies; thoraco-lumbar spine
MeSH Terms: conditions — Disease | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): patients with degenerative pathology of the thoraco-lumbar-sacral spine
  Interventions: Other: screening

INTERVENTIONS:
Other: screening — Comprehensive screening of bone metabolic status and bone fragility in the largest cohort to date of patients with degenerative spinal diseases

SUMMARY:
The present study is related to the project "ORTHOSPINE FITNESS: WHICH MARKERS OF MUSCULOSKELETAL HEALTH CAN EXPLAIN COMPLICATIONS IN SPINE SURGERY?", winner of the Ministry of Health Call, financed by the European Union, "M6/C2_CALL 2023", Project Code " PNRR- MCNT2-2023-12378098", Call section "Non-chronic chronic diseases transmissible diseases (MCnT2) with a high impact on health systems".

Complications of spinal surgery still represent a significant and unsolved problem. Their incidence is between 7 and 20%, with a high percentage of mechanical complications observed in patients operated on for degenerative pathologies. Readmissions, re-operations and subsequent rehabilitation treatments have a heavy impact on patients and the entire healthcare system.

DETAILED DESCRIPTION:
The study proposed, financed through the "PNRR-MCNT2-2023-12378098" call, is a multicenter study on a large cohort of patients undergoing spinal surgery for degenerative pathologies of the thoraco-lumbar spine, which has as its general objective to establish a comprehensive preoperative screening of bone health and the musculoskeletal system, combining advanced imaging and modeling (HRpQCT images of bone microstructure at peripheral sites and related computational assessment of bone mechanical properties), assessment of physical fragility (including muscle strength and assessment of proprioception/fall risk), cellular and molecular analyzes of bone fitness and bone-muscle cross-talk, and assessment of nutritional status.

The results of the project will allow us to: (i) define a concept of "surgical suitability" to evaluate patients candidates for elective spinal surgery and possibly improve the surgical decision-making process (for example the choice of fixation and instrumentation); (ii) identify a minimum set of significant and independent markers to monitor in future interventional studies aimed at reducing the risk of adverse events in spinal surgery, (iii) allow patient-specific preoperative interventions (such as nutritional supplementation, physical pre-habilitation or administration of bone anabolic agents)

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years;
* diagnosis of degenerative pathology of the spinal column of the thoraco-lumbo-sacral tract;
* patients candidates for surgical treatment for the aforementioned pathology during the study period;
* willingness to participate in the study and sign the specific informed consent

Exclusion Criteria:

* presence of tumors or infections in the spinal column;
* presence of degenerative pathology of the spine without surgical indication;
* presence of degenerative pathology of the spinal column at the cervical level.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
radiological images | at baseline (day 0)
  constructed mechanical models from HR-pQCT data to quantify mechanical stiffness and bone strength at peripheral sites, which have already been shown to be effective predictors of fractures independent of DXA, and attempted their association with adverse events monitored during the follow-up
biological samples | at baseline (day 0), after 6 months, after 12 months
  The biopsies will be analyzed for analyzes at the level of secreted proteins (secretome) and gene expression. The bone harvest will be waste material obtained from the laminectomy, while the muscle harvest will be carried out in very small quantities from the posterior paravertebral muscles
pain | at baseline (day 0), after 12 months
  Pre-operative baseline assessment of pain level will be performed by self-administering validated questionnaires with the visual analogue scale (0-10)
Quality of life | at baseline (day 0), after 6 months, after 12 months
  the quality of life of the patients will be tracked by questionnairs
nutritional informations | since day 1 to day 14
  administration of a questionnaire to patients food frequency (Food Frequency Questionnaire - FFQ), which is an accurate measurement of nutrient intake within a 14-day period, using a diary food.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Istituto Ortopedico Rizzoli, Bologna
  - Azienda ospedaliera universitaria Luigi Vanvitelli, Napoli

IPD SHARING:
Plan to Share IPD: Undecided